CLINICAL TRIAL: NCT04604210
Title: A Pilot Randomized Trial of Distinct Symptom-specific Targets for Transcranial Magnetic Stimulation in Patients With Depression and Anxiety
Brief Title: Symptom-specific TMS Targets for Depression and Anxiety
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Shan Siddiqi, MD, Assistant Professor, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2020P002296
Record Dates: First submitted 2020-10-16; First posted 2020-10-27 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Depression; Anxiety; Major Depressive Disorder
Keywords: TMS; Transcranial; Neuromodulation; Brain stimulation; Depression; Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders; Depressive Disorder, Major | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Parallel-group double-blind randomized, controlled trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants will be blinded to which target is expected to improve which symptom.
  Study investigators (with the exception of the treatment administrator), including the outcomes assessor, will be blinded to which participant is receiving which treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Dysphoric target (Experimental): The "dysphoric" target is a region in the dorsolateral prefrontal cortex. TMS targeted to this region has been shown to be more effective for depression than anxiety.
  Interventions: Procedure: Transcranial magnetic stimulation
- Anxiosomatic target (Experimental): The "anxiosomatic" target is a region in the dorsomedial prefrontal cortex. TMS targeted to this region has been shown to be more effective for anxiety than depression.
  Interventions: Procedure: Transcranial magnetic stimulation

INTERVENTIONS:
Procedure: Transcranial magnetic stimulation — Transcranial magnetic stimulation (TMS) is a noninvasive FDA-approved technique that is commonly used as a treatment for depression. It has been shown to focally activate specific brain regions that are believed to be underactive in patients suffering from depression. In this study, TMS will be administered within FDA-approved guidelines under the supervision of a physician with experience in administering the treatment and monitoring for complications.
  Other Names: TMS

SUMMARY:
This pilot study aims to compare two different treatment targets for transcranial magnetic stimulation, an FDA-approved treatment for major depressive disorder (MDD), in terms of their relative efficacy for depression versus anxiety.

DETAILED DESCRIPTION:
Transcranial magnetic stimulation (TMS) is a safe, noninvasive FDA-cleared technique that is commonly used as a treatment for MDD. It has been shown to focally activate specific brain regions that are believed to be underactive in these patients. This study aims to compare two different TMS targets in the prefrontal cortex. TMS will be administered within FDA-approved guidelines under the supervision of a physician with experience in administering the treatment and monitoring for complications.

This will be a prospective double-blind randomized controlled trial to assess the comparative efficacy of two different TMS targets within the prefrontal cortex (PFC). The "dysphoric" target in the dorsolateral PFC is believed to be more effective for depression, while the "anxiosomatic" target in the dorsomedial PFC is believed to be more effective for anxiety.

Patients with comorbid depression and anxiety will receive 6 weeks of TMS following standard clinical parameters (30 treatments over 6 weeks, 10 Hz frequency, 3000 pulses) with MRI-guided neuronavigation. Participants will be randomized to either the dysphoric or anxiosomatic target. Both targets are believed to be effective treatments for this patient population. Participants and raters will remain blinded to the group assignment. All participants will receive resting-state functional MRI scans before and after the course of treatment in order to study physiological changes.

The dysphoric target is expected to induce greater relative improvement in depression, while the anxiosomatic target is expected to induce greater relative improvement in anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18 to 65
* Meeting FDA guidelines for clinical TMS (DSM-5 diagnosis of major depressive disorder with at least one failed antidepressant trial)1
* Beck Depression Inventory (BDI) score of 20 or higher
* Beck Anxiety Inventory (BAI) score of 16 or higher

Exclusion Criteria:

* History of:

  * Moderate or severe substance use disorder in the past six months as defined by DSM-5 criteria, with the exception of cannabis and nicotine use disorders.
  * Dementia, as defined by treating neurologist
  * Moderate or severe autism spectrum disorder
  * Bipolar disorder
  * Schizophrenia spectrum disorders
* Current evidence of:

  * Substance-induced mood disorder
  * Active psychotic symptoms
  * Active suicidal ideation
* Contraindications to rTMS treatment:

  * Seizure disorder
  * Significantly elevated seizure risk, as determined by clinician assessment
  * Presence of metallic objects within the head
  * Presence of an implanted neurostimulation device within the head
* Contraindications to MRI

  * Severe claustrophobia
  * Severe pain/illness exacerbated by lying prone in the scanner
  * Presence of non-MRI compatible metal foreign bodies or implants
  * Weight in excess of 350 lbs
  * Shoulder width in excess of maximum tolerable width for scanner

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-02-03 (Actual); Primary Completion 2023-12-28 (Actual); Study Completion 2023-12-28 (Actual)

PRIMARY OUTCOMES:
Beck Anxiety Inventory (BAI) | Baseline (before treatment), 3 weeks (after 15 treatments), and 6 weeks (after 30 treatments)
  The primary outcome will be the rank-transformed ratio of BDI change to BAI change
Beck Depression Inventory (BDI) | Baseline (before treatment), 3 weeks (after 15 treatments), and 6 weeks (after 30 treatments)
  The primary outcome will be the rank-transformed ratio of BDI change to BAI change

SECONDARY OUTCOMES:
Resting-state functional MRI (rsfMRI) scan | Baseline (before treatment) and 6 weeks (after 30 treatments)
  Functional MRI scan will be conducted before and after treatment in order to assess for treatment-induced changes in brain connectivity
Temperament and Character Inventory, Revised 140-item (TCI-R 140) | Baseline (before treatment) and 6 weeks (after 30 treatments)
  Psychobiologically-based personality inventory which measures seven personality dimensions (harm avoidance, novelty seeking, reward dependence, persistence, self-directedness, cooperativeness, and persistence). For each dimension, this yields a scaled T-score (mean score of 50 with standard deviation of 10). This is an overall estimate of personality traits, and there are no "better" or "worse" traits.
NIH Toolbox cognitive battery | Baseline (before treatment) and 6 weeks (after 30 treatments)
  An interactive computerized battery of cognitive tasks which is used to compute an overall index of crystallized and fluid cognition. For each cognitive subscale, this yields a scaled T-score (mean score of 100 with standard deviation of 10).
Multidimensional task-based emotional assessment | Baseline (before treatment) and 6 weeks (after 30 treatments)
  An interactive computerized battery of emotional tasks, including Aversion-Reward Conflict, Emotion Conflict Resolution, Multiple Source Interference, Fear Conditioning/Extinction, Gambling, and Associative Learning Tasks. Each task will yield results for accuracy and reaction time.
Pain at the stimulation site | Baseline (before treatment) and 6 weeks (after 30 treatments)
  Participants will be asked to rate treatment-induced pain/discomfort on a scale of 1 to 10
Multidimensional battery of emotional questionnaires | Baseline (before treatment) and 6 weeks (after 30 treatments)
  A computerized battery of questionnaires including the Anxiety Sensitivity Index, Adult Temperament Questionnaire, Emotion Reactivity Scale, Barratt Impulsivity Scale, Adult ADHD Self-Rating Scale, Brief Inventory of Executive Functioning. Each scale yields a raw score.

CONTACTS AND LOCATIONS:
Overall Officials: Shan H Siddiqi, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham & Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided
De-identified survey response data and/or neuroimaging data may be shared with collaborators for further analysis.